CLINICAL TRIAL: NCT06386952
Title: To Compare People With T2DM Who Have Double Dorsal Cervical Fat (Double Hump) Versus Who do Not Have Double Dorsal Cervical Fat (Double Hump)
Brief Title: To Compare People With T2DM Who Have Double Hump Versus Who do Not Have Double Hump
Status: Recruiting | Type: Observational
Sponsor: Diabetes Foundation, India (Other)
Collaborators: National Diabetes Obesity and Cholesterol Foundation (Other)
Responsible Party: Principal Investigator, Dr Anoop Misra, Director, Diabetes Foundation, India
Other Study IDs: 02/2024-2025
Record Dates: First submitted 2024-04-20; First posted 2024-04-26 (Actual); Last update posted 2024-04-26 (Actual); Status verified 2024-04

CONDITIONS: Type 2 Diabetes Mellitus With Complication

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- With Double Dorsal Cervical Fat: T2DM with Double Dorsal Cervical Fat (Double Hump)
- Without Double Dorsal Cervical Fat: T2DM without Double Dorsal Cervical Fat (Double Hump)

SUMMARY:
Hypothesis: Double Hump in people with T2D is associated with higher magnitude of complication than people with single hump or no hump

Objectives: To correlate single and double hump with diabetes complication T2DM patient will be recruited from endocrine OPD

1. Clinical History and Examination:

1. General Physical Examination: Height, weight, waist circumference, hip circumference, BMI, Blood Pressure, Hand grip. Buffalo Hump.
2. Complications Assessment: Patient will be analyzed for:

Micro Vascular

(a) Diabetic retinopathy (i) Mild NPDR (ii) Mod NPDR (iii) Macular Edema / CSME (b) Neuropathy (Mild/Mod/Severe) (c) Chronic Kidney Disease (i) Micro/Macro albumin urea (ii) Increased Creatinine (iii) Decreased eGFR

Macro Vascular

1. Low ABI/PAD
2. CVD-MI/PTCA/CABG/Heart Failure
3. CVS-Stroke/ TIA/Carotid Blockage >50%

DETAILED DESCRIPTION:
The development of type 2 diabetes mellitus (T2DM) as a major public health problem in Asian Indians. Asian Indians develop T2DM at a younger age, and progresses faster than in other ethnic groups. As a result, many diabetes complications are more prevalent and in more advanced stages in Asian countries than in other regions. Asian Indians have one of the highest incidence rates of pre-diabetes and T2DM among all major ethnic groups, and the conversion from pre-diabetes to T2DM occurs more rapidly in this population. According to the Indian Council of Medical Research- India diabetes study (57 117 individuals), the prevalence of prediabetes in all 15 states was 7·3%.

The tendency of Asian Indian to develop T2DM is enhanced by greater insulin resistance, dysglycemia, subclinical inflammation and non-alcoholic fatty liver disease (NAFLD).

"Buffalo hump," or a dorso cervical fat pad, is a term that refers to a collection of excess fat behind the neck that causes the shoulders to develop a hump-like shape. It can be caused by a variety of underlying conditions or medications.

A buffalo hump is most commonly a result of Cushing syndrome, a disorder of excess cortisol, a naturally occurring hormone that is involved in a variety of bodily processes, such as metabolism. High levels of the hormone cortisol can lead to increased fat synthesis. With Cushing syndrome, the fat produced often deposits in the neck, known as lipodystrophy. This produces the characteristic buffalo hump. Cushing syndrome may be caused by an adrenal tumor, lung tumor, or glucocorticoid medications. If Cushing syndrome is caused by a pituitary tumor, it is known as Cushing disease.

This Prospective observational study will be of 12 months' duration where 100 T2DM patients from urban areas of Delhi will be randomly screened. The population will be representative of different socio-economic strata of the society. Clinical and dietary profiles, blood pressure and phenotypic markers (acanthosis nigricans, buffalo hump, skin tags: xanthelasma, double chin, arcus, hirsutism and tendon xanthoma), diabetic retinopathy, peripheral arterial disease (PAD), neuropathy, nephropathy HTN, CHF, CT Coronary Angiography, CAD, Arrhythmias, Coronary Calcification, Cerebrovascular Disease, peripheral vascular disease, micro albumin urea, fibro scan and hand grip (average of three values) JAMAR measurement will be assessed.

To diagnose a buffalo hump and its underlying cause, a healthcare professional generally will review the individual's current medications and medical history, as well as conduct a physical examination.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with T2DM (up to 30 years Duration)
2. Age 20 to 70 years
3. BMI >25 kg/m² to >40 kg/m²
4. Gender- Both (Male & Female)

Exclusion Criteria:

1. Alcoholic with Moderate to Severe.
2. BMI >40 kg/m²
3. Congestive heart disease
4. Positive hepatitis B or hepatitis C, secondary causes of fatty liver (eg. consumption of amiodarone and tamoxifen) and congestive hepatopathy.
5. Severe end organ damage or chronic diseases: renal/hepatic failure, any malignancy, major systemic illness etc.

Ages: 20 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patient with T2DM visiting Fortis CDOC Hospital will be enrolled in 2 groups cases and controls.
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2024-05-01 (Estimated); Primary Completion 2025-05-31 (Estimated); Study Completion 2025-06-30 (Estimated)

PRIMARY OUTCOMES:
Double Hump increases diabetes complications | 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Anoop Misra, MD, Principal Investigator — National Diabetes Obesity and Cholesterol Foundation
Locations (1):
- Anoop misra, New Delhi, National Capital Territory of Delhi, India

IPD SHARING:
Plan to Share IPD: No